CLINICAL TRIAL: NCT07230535
Title: A Randomised Control Trial Evaluating Well Being and Patient Reported Outcomes After Open vs Robotic Single-port Nipple Sparing Mastectomy With DIEP Reconstruction
Brief Title: Evaluation of Wellbeing and Patient Reported Outcomes After Open vs Robotic Mastectomy With DIEP Reconstruction
Acronym: REBORN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Arnold Hill, Professor, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25/56
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer, Breast Neoplasms; Breast Reconstruction; DIEP Flap Breast Reconstruction; Robotic Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Assisted Nipple Sparing Mastectomy (Experimental): Participants randomised to this arm will undergo robotic-assisted nipple-sparing mastectomy using a single-port robotic platform. Surgery will be performed via a single axillary incision. Immediate breast reconstruction will be undertaken according to the pre-specified reconstruction plan:
  Implant-based reconstruction or Autologous deep inferior epigastric perforator (DIEP) flap reconstruction
  Robotic-assisted procedures will be delivered at the designated network hub hospital.
  Interventions: Procedure: Robotic Assisted Nipple Sparing Mastectomy
- Standard Open Nipple Sparing Mastectomy (Active Comparator): Participants randomised to this arm will undergo standard open nipple-sparing mastectomy performed via a conventional incision in accordance with institutional practice. Immediate breast reconstruction will be undertaken according to the pre-specified reconstruction plan:
  Implant-based reconstruction or Autologous deep inferior epigastric perforator (DIEP) flap reconstruction
  Standard open procedures will be performed either at the referring network site or centrally, depending on reconstructive requirements.
  Interventions: Procedure: Standarding Open Nipple Sparing Mastectomy

INTERVENTIONS:
Procedure: Robotic Assisted Nipple Sparing Mastectomy — Description: Nipple-sparing mastectomy performed using a single-port robotic surgical system through a single axillary incision, preserving the nipple-areolar complex where oncologically appropriate.
  Arms: Robotic Assisted Nipple Sparing Mastectomy
Procedure: Standarding Open Nipple Sparing Mastectomy — Nipple-sparing mastectomy performed using an open surgical approach through a conventional incision, preserving the nipple-areolar complex where oncologically appropriate.
  Arms: Standard Open Nipple Sparing Mastectomy

SUMMARY:
Nipple-sparing mastectomy (NSM) preserves the nipple-areolar complex (NAC) and is associated with improved cosmetic outcomes, body image, and patient satisfaction compared with more ablative techniques. Its use has expanded in both therapeutic and risk-reducing settings, including ductal carcinoma in situ (DCIS) and early-stage invasive breast cancer, where the NAC is not clinically or radiologically involved. Multiple observational and cohort studies support the oncological safety of NSM in appropriately selected patients, provided meticulous surgical technique and pathological assessment are employed to minimise the risk of residual disease.

Robotic-assisted NSM has emerged as a minimally invasive alternative to conventional open techniques. Robotic platforms offer enhanced three-dimensional visualisation, improved instrument articulation, and ergonomic advantages that may facilitate precise dissection while reducing surgeon fatigue. Single-port robotic systems enable NSM to be performed through a single axillary incision, potentially reducing visible scarring and postoperative discomfort while maintaining oncological principles. Early series from high-volume centres have demonstrated the technical feasibility and short-term safety of robotic NSM, with outcomes broadly comparable to open NSM and signals of potential aesthetic benefit. However, these data are largely non-randomised and derived from single-centre experiences.

Despite the increasing adoption of both conventional and robotic NSM, there remains a paucity of high-quality prospective evidence evaluating patient-reported outcomes (PROs). Validated instruments such as the Breast-Q, Hopwood Body Image Scale, and Aesthetic Item Scale (AIS) provide robust measures of patient satisfaction, psychosocial well-being, and aesthetic outcome, yet randomised comparisons of robotic versus open NSM using these tools are lacking. In particular, there is limited evidence examining whether the proposed cosmetic and experiential advantages of robotic surgery translate into meaningful improvements in PROs across different reconstructive pathways.

Breast reconstruction is a critical determinant of postoperative quality of life following mastectomy. Both implant-based reconstruction and autologous reconstruction using deep inferior epigastric perforator (DIEP) flaps are established techniques, each with distinct risk profiles, recovery trajectories, and long-term outcomes. Autologous DIEP reconstruction is associated with superior long-term satisfaction and physical well-being in many patients, while implant-based reconstruction remains the most commonly performed approach nationally. Evaluating NSM techniques across both reconstructive modalities enhances the generalisability and clinical relevance of trial findings.

The REBORN Network Trial is a multicentre, randomised controlled study conducted within an Irish cancer network using a hub-and-spoke model for robotic surgery delivery. Patients undergoing mastectomy with immediate reconstruction are stratified by reconstruction type (implant-based or DIEP flap) and randomised to receive either robotic-assisted or conventional open NSM. Robotic procedures are centralised within a designated surgical hub, while open procedures are delivered either locally or centrally, depending on reconstructive requirements. This design enables equitable access to robotic surgery while maintaining oncological safety and surgical expertise.

By comparing robotic-assisted and open NSM within both implant and DIEP reconstruction cohorts using validated PRO measures, this study aims to determine whether robotic technology confers measurable benefits in patient satisfaction, body image, and aesthetic outcome. The findings will inform patient counselling, surgical decision-making, and future service development within networked breast cancer care systems.

DETAILED DESCRIPTION:
The study will be a prospective, multicentre, single-blinded (outcome assessor-blinded), randomised controlled trial conducted within an Irish cancer network using a hub-and-spoke model for robotic surgery delivery. The trial will compare robotic-assisted versus conventional open nipple-sparing mastectomy (NSM) in patients undergoing immediate breast reconstruction.

Participants will be stratified by type of reconstruction and randomised in a 1:1 ratio within each stratum. Two reconstruction cohorts will be studied:

Implant Reconstruction Cohort Arm A1: Robotic-assisted NSM with immediate implant-based reconstruction Arm A2: Standard open NSM with immediate implant-based reconstruction

Autologous Reconstruction (DIEP) Cohort

Arm B1: Robotic-assisted NSM with immediate DIEP flap reconstruction Arm B2: Standard open NSM with immediate DIEP flap reconstruction

Randomisation will be stratified by recruiting site and reconstruction type. Robotic-assisted NSM procedures will be performed at the designated network hub, while standard open NSM procedures will be undertaken either at the referring site or centrally, depending on reconstructive requirements.

All patients eligible for mastectomy and immediate reconstruction will be screened for inclusion. Eligibility for nipple-sparing mastectomy will be determined based on clinical and radiological criteria, including the absence of tumour involvement of the skin or nipple-areolar complex and an adequate tumour-to-nipple distance, in accordance with institutional and national guidelines. Patients not suitable for NSM will not be randomised and will undergo standard-of-care mastectomy outside the trial.

Blinding will be applied to outcome assessment. Independent assessors evaluating aesthetic outcomes and analysing patient-reported outcome measures, including Breast-Q, Hopwood Body Image Scale, and Aesthetic Item Scale (AIS), will be blinded to treatment allocation. Due to the nature of the surgical interventions, blinding of patients and surgeons will not be feasible.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Candidates who have already been selected to undergo mastectomy (of any kind) and immediate DIEP reconstruction by the breast MDT for the following indications:

  1. Genetic mutation carriers undergoing risk-reducing mastectomy.
  2. Ductal carcinoma in situ (DCIS) requiring mastectomy.
  3. Early invasive breast cancer requiring mastectomy.
  4. For those considered for Nipple Sparing Mastectomy randomisation arms the tumour must not have skin involvement and no evidence of invasive disease within 1cm of skin, nipple or Pec major muscle (as proven on MRI).
* Candidates for immediate breast reconstruction with DIEP reconstruction
* Fluent in English
* Fit for general anaesthetic
* Signed informed consent form

Exclusion Criteria:

* Advanced breast cancer with skin involvement for Nipple Sparing Mastectomy Arms
* Nipple involvement for Nipple Sparing Mastectomy Arms.
* Prior chest wall radiation therapy
* Pregnancy
* Lactation
* Patients with insufficient English to sign an informed consent (i.e. interpreter required).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the difference in patient-reported outcomes at 12 months postoperatively. | Up to 12 months post operative
  Difference in patient-reported outcomes at 12 months postoperatively, assessed using the BREAST-Q Reconstruction Module

CONTACTS AND LOCATIONS:
Locations (1):
- Beaumont RCSI Cancer Centre, Beaumont, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and anonymised data related to the results will be made available through peer review publication.
Supporting Information: Study Protocol
Access Criteria: Peer review publications

REFERENCES:
- [Background] Toesca A, Sangalli C, Maisonneuve P, Massari G, Girardi A, Baker JL, Lissidini G, Invento A, Farante G, Corso G, Rietjens M, Peradze N, Gottardi A, Magnoni F, Bottiglieri L, Lazzeroni M, Montagna E, Labo P, Orecchia R, Galimberti V, Intra M, Sacchini V, Veronesi P. A Randomized Trial of Robotic Mastectomy Versus Open Surgery in Women With Breast Cancer or BrCA Mutation. Ann Surg. 2022 Jul 1;276(1):11-19. doi: 10.1097/SLA.0000000000004969. Epub 2021 Jun 9. PMID 34597010